CLINICAL TRIAL: NCT02223546
Title: Pilotstudy: Diurnal Changes in Choroidal Volume
Brief Title: Circadian Macular Volume Changes in the Choroid
Acronym: CVdi
Status: Completed | Type: Observational
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Other Study IDs: CVdi
Record Dates: First submitted 2014-08-21; First posted 2014-08-22 (Estimated); Results first posted 2020-09-24 (Actual); Last update posted 2020-09-24 (Actual); Status verified 2020-09

CONDITIONS: Choroid Physiology

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- healthy subject: healthy subject, every 3 hour measurement

SUMMARY:
Choroidal volume measured fluctuates significantly over a 24 hour time frame.

DETAILED DESCRIPTION:
All patients undergo enhanced depth imaging (EDI) by the Spectralis SD-OCT device (Heidelberg Spectralis HRA2, Heidelberg Engineering, Heidelberg, Germany). SD-OCT measurements will be performed in both eyes after pupil dilation.

Scanning Protocol: This studies choroidal volume measurement protocol has been previously published. In short, 31 high resolution B-scans centered at the fovea will be obtained by a single investigator. To optimize image quality each B-scan will be averaged from at least 25 individual scans using the build in eye tracking software (TrueTrack, Heidelberg Engineering, Heidelberg, Germany). Scan length will be set to 9.3mm and spacing to 240µm, resulting in a 30x25 degree area around the fovea.

Each individual will undergo SD-OCT measurement every 3 hours within a 24 hour timeframe (at 0, 3, 6, 9 12, 15, 18, and 21 o'clock; 8 times total). Additionally, automated blood pressure measurement and Goldmann applanation tonometry will be performed every 3 hours. Subject will be instructed to sleep in erect position from 21 to 6 o'clock, and will be awoken for examination at 0 and 3.

OCT Analysis: Two retinal specialists will manually adjust the segmentation lines for automated choroidal volume calculation by the devices build in software. Choroidal thickness is defined as the layer between the outer boarder of the retinal pigment epithelium (RPE) and the hyper reflective layer behind the large vessels of the choroid (chorio-scleral interface). The devices Software thus generates a three-dimensional choroidal thickness map, divided according to the Early Treatment Diabetic Retinopathy Study (EDTRS) grid. In addition to this, subfoveal choroidal thickness will be measured manually using the SD-OCTs integrated caliper tool, drawing a perpendicular line to the RPE within the aforementioned bounds.

This is considered a pilot study, so explorative data analysis will be performed.

ELIGIBILITY:
Inclusion Criteria:

* age 18-65, signed informed consent form,

Exclusion Criteria:

* any ocular pathology, including history of ocular surgery or trauma, use of ocular medication, elevated intraocular pressure (IOP), or significant vitreous floaters. Further exclusion criteria were current use of any systemic medications, history of cardio-vascular disease, diabetes mellitus, or hypertension

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Helathy human subjects
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2013-10; Primary Completion 2014-01 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gerald Seidel, MD, Principal Investigator — Medical University of Graz
Locations (1):
- Department of Ophthalmology, Medical University of Graz, Graz, Styria, Austria

REFERENCES:
- See also: PMID 25447108 — https://www.ncbi.nlm.nih.gov/pubmed/25447108

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Healthy Subject
Started | 15
Completed | 15
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Healthy Subject
Number analyzed (Participants) | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 26 (1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 8

OUTCOME MEASURES:

1. Primary Outcome: Macular Choroidal Volume
Description: macular choroidal volume in the central 6mm
Time Frame: daily average out of measurements every 3 hours within a 24 hour timeframe
Measure: Mean (Standard Deviation); unit: mm^3
Arm/Group | Healthy Subject
Number analyzed (Participants) | 15
mm^3 | 10.33 (2.53)

2. Secondary Outcome: Subfoveal Choroidal Thickness
Time Frame: daily average out of measurements every 3 hours within a 24 hour timeframe
Measure: Mean (Standard Deviation); unit: µm
Arm/Group | Healthy Subject
Number analyzed (Participants) | 15
µm | 378.1 (111.3)

3. Other Pre Specified Outcome: Mean Ocular Perfusion Pressure
Description: mean arterial pressure (MAP) is defined as DBP + 1/3(SBP - DBP); mean ocular perfusion pressure results from 2/3(MAP - IOP).
Time Frame: every 3 hours within a 24 hour timeframe
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Healthy Subject
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes